CLINICAL TRIAL: NCT06576063
Title: Effects of the Regular Use of Antibacterial Photodynamic Therapy as an Adjunctive Treatment on Oral Hygiene in Elderly Persons Living at Home or at Care Homes
Brief Title: Antibacterial Photodynamic Therapy as an Adjunctive Treatment on Oral Hygiene in Elderly Persons
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koite Health Oy (Industry)
Collaborators: University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LumoKoti2024
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Dental Plaque; Bleeding of Subgingival Space; Oral Complication
Keywords: Lumoral; Preventive oral care; Antibacterial photodynamic therapy (aBPT); aMMP-8; Plaque control; Oral hygiene
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: Randomized clinical study on a medical device.
Who Masked: Outcomes Assessor
Masking Description: Data will be collected using individual study codes for participants. Study codes do not reveal which group the participant has belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Standard oral hygiene methods and adjuvant use of Lumoral Treatment device
  Interventions: Device: Lumoral Treatment; Behavioral: Standard oral hygiene methods
- Control group (Active Comparator): Standard oral hygiene methods
  Interventions: Behavioral: Standard oral hygiene methods

INTERVENTIONS:
Device: Lumoral Treatment — Home-use of photodynamic antibacterial dual-light device, used with a marker substance (indocyanine green)
  Arms: Study group
Behavioral: Standard oral hygiene methods — Best available standard oral self-care hygiene methods performed at home and instructed by oral healthcare professionals, supported by professional cleaning at the oral healthcare clinic

SUMMARY:
On average, the dental condition of elderly people is poor due to various reasons. The importance of oral health maintenance of the ageing population has been recognized by the World Health Organization (WHO), as oral health plays a key role in reaching the global goal of the "Decade of Healthy Ageing 2021-2030".

New measures for maintaining good oral health are welcome. The use of antibacterial photodynamic therapy (aPDT) and antibacterial blue light (aBL) has been studied and found to reduce the amount of plaque in the mouth. The Lumoral device is a CE-marked home medical device combining aPDT and aBL, and it is effective in reducing the development of plaque and harmful bacteria in the plaque. The device has also been shown to be easy and safe to use. In this study, a combination of regular dental appointments with the importance of enhanced dental self-care, will be tested as one regional solution for reaching the global goal set by WHO.

DETAILED DESCRIPTION:
The ageing population is increasing rapidly worldwide. In the year 2000, there were 69 million people over the age of 80 in the world, and it is estimated that by the year 2030, 1 out of 6 persons will be 60 years of age or more worldwide. The proportion of the ageing population having their natural teeth left is also increasing. In Finland, the average number of toothless people aged over 65 has decreased from 44% measured in the year 2000 to 21% in 2011.

As people get older, their ability to function deteriorates, and the elderly, especially those living in round-the-clock care, have been found to have shortcomings in maintaining oral hygiene. Toothlessness is reduced in the elderly population living in care homes, too. According to a Study in Finland, in 2003, 52 % of inhabitants were toothless in enhanced service housing, and in 2017, the proportion of toothless had decreased to 38%. In 2017-2018, inhabitants of elderly care homes had an average of 13.8 teeth. Only a small proportion of the population had clean teeth, and the worse the level of oral hygiene, the worse the quality of life.

The World Health Organization has proposed a "Decade of Healthy Ageing 2021-2030" action plan to encourage countries to develop and implement policies and programs to promote healthy ageing and improve the quality of life in the older population. While there is an interrelation between oral and systemic health, periodontal health has been linked to several chronic systemic conditions such as diabetes and cardiovascular diseases via shared inflammatory pathways. Good oral health enables daily functions like eating and speaking, while tooth loss, hyposalivation and other oral conditions obstruct oral functions and make nutritional intake more difficult. Bad oral condition also affects social interaction and quality of life. As oral functioning declines, it is associated with a decline in general function and weakness in the older population, and it can eventually lead even to disability and loss of independence. Therefore, the World Health Organization together with the World Dental Federation have recognized the importance of oral health maintenance and functioning to enable healthy ageing in older adults.

The dental condition of elderly persons is often poor. Cavities and dental connective tissue disease are relatively common in persons of 75 and older. Untreated oral infections predispose elderly people to pneumonia, among other complications. Chronic oral infectious diseases, and sometimes fatal complications, are preventable with good oral hygiene. Regular cleaning of the mouth and teeth from plaque is still the most important thing for keeping the mouth healthy. One third of the aged population in Finland suffers from dry mouth due to various illnesses or the use of many medications. Lack or reduction of saliva may predispose to inflammatory diseases in the mouth. If multiple medications are in use simultaneously, the dry mouth symptoms may even worsen.

The use of antibacterial photodynamic therapy (aPDT) and antibacterial blue light, as adjunctive treatments to standard oral home care has been studied and found to reduce the amount of plaque in the mouth. The Lumoral device is a CE class IIa -marked medical device for home use that has been found to be effective in reducing the development of plaque and harmful bacteria in the plaque. The performance of the device is based on the aPDT method, in which the photosensitive substance in the Lumorinse mouthwash attaches to the bacterial coating and is activated as an antibacterial by light. The antibacterial effect is applied directly to the plaque, reducing the impact on the normal oral flora. Preliminary studies have found that the method reduces inflammatory factors in periodontitis. In addition, the heat produced by the device also enhances saliva production, which also affects maintaining good oral health. Unpublished data from a randomized clinical trial conducted by the University of Helsinki in which Lumoral was used by the residents of elderly 24-hour care also showed that the device was safe to use, and it had a significant impact on oral health measured by the Community Periodontal Index.

This study aims to determine the effectiveness of the Lumoral Treatment method as an adjunctive treatment on oral hygiene, inflammatory load, and dryness of mouth in elderly people living at home or at care homes, and who are regular customers with the study sites.

ELIGIBILITY:
Inclusion Criteria:

* An elderly (age ≥ 65 years) person living at home or at care home, with a possibility to regular dental care appointments
* Ability to understand and sign the informed consent
* At least 10 teeth in the mouth, including implants
* Ability to understand and follow the study protocol, including tooth brushing and following the instructions for the use of Lumoral Treatment, based on the assessment of the investigator

Exclusion Criteria:

* Uncontrolled diabetes mellitus (DM)
* Severe dementia or other similar conditions that may restrict understanding of the study information and protocol
* Presence of any physical limitation or restriction that might restrict Lumoral use
* Active smoking and use of other tobacco products
* Use of antibiotics within 4 weeks week prior study
* Oral thrush
* Known sensitivity to near-infrared or antibacterial blue light.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing (BOP) | 9 months
  Change in the inflammatory parameter BOP.A full-mouth assessment at six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual). Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus. Dichotomous scoring to each site of the tooth as bleeding "1 present" and "0 absent". BOP is reported as the percentage (%) of sites with positive findings.
  Calculation formula: number of bleeding sites/ 6 times number of teeth.

SECONDARY OUTCOMES:
Plaque index (RMNPI) | 9 months
  Assessment of six index teeth, measured at four sites per tooth
  * Dichotomous scoring to each site of the tooth as plaque "1 present" and "0 absent"
  * RMNPI reported as the percentage (%) of sites with plaque
  * Calculation formula: number of sites with plaque/ 4 times number of teeth
Periodontal Pocket Depth (PPD) | 9 months
  A full-mouth assessment, measured at six sites per tooth. Assessed from the base of the pocket to the gingival margin (mm)
Active matrix metalloproteinase 8 (aMMP-8) | 9 months
  Change in periodontal inflammation marker aMMP-8. The oral rinse fluid sample collection and the aMMP-8 marker analysis will be performed using Periosafe test (Dentognostics GmbH) according to the manufacturer's instructions.
Oral Bacterial flora | 9 months
  Quantification of periodontopathic bacteria by 16S rRNA sequencing analysis
  - Microbiological samples can be collected using Iso Taper Paper Points, size-20 (VDW GmbH) from selected gingival/periodontal pockets with maximum initial probing depth. The paper points can be placed into sterile, small-aliquot containers, and immediately stored at -20°C until analysis
Dryness of Mouth (DOM) | 9 months
  Clinical, visual assessment of oral mucosal moisture/dryness:
  0 points: Saliva secretion appears normal (saliva serous, runny)
  1. point: Oral mucosa shiny and tight; and/or saliva foamy or mucousy; and or only a little clear saliva at the bottom of mouth
  2. points: Mouth completely dry, mirror sticks to cheek or tongue, mucous membranes often reddened; and/or knuckles on the surface of the tongue have disappeared; and/or mouth appears carstic
OHIP-14 questionnaire | 9 months
  Measures people's perception of the social impact of oral disorders on their well-being.
  Fourteen items of OHIP are divided into seven dimensions: functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability, and handicaps. Responses are made on a 5-point scale (from 0 = never, to 4 = very often).
Adverse events | 9 months
  Any suspicion of an adverse event related to the investigational device, the treatment method, or the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Timo Sorsa, Professor, Principal Investigator — University of Helsinki
Locations (3):
- Finland (3):
  - SuperSuu, Loviisa, Uusimaa
  - SuperSuu, Sipoo, Uusimaa
  - KotiHammas, Vantaa, Uusimaa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cugini M, Thompson M, Warren PR. Correlations between two plaque indices in assessment of toothbrush effectiveness. J Contemp Dent Pract. 2006 Nov 1;7(5):1-9. PMID 17091134
- [Background] Lahteenmaki H, Patila T, Raisanen IT, Kankuri E, Tervahartiala T, Sorsa T. Repeated Home-Applied Dual-Light Antibacterial Photodynamic Therapy Can Reduce Plaque Burden, Inflammation, and aMMP-8 in Peri-Implant Disease-A Pilot Study. Curr Issues Mol Biol. 2022 Mar 8;44(3):1273-1283. doi: 10.3390/cimb44030085. PMID 35723308
- [Background] Nikinmaa S, Moilanen N, Sorsa T, Rantala J, Alapulli H, Kotiranta A, Auvinen P, Kankuri E, Meurman JH, Patila T. Indocyanine Green-Assisted and LED-Light-Activated Antibacterial Photodynamic Therapy Reduces Dental Plaque. Dent J (Basel). 2021 May 3;9(5):52. doi: 10.3390/dj9050052. PMID 34063662
- [Background] Saarela RKT, Hiltunen K, Mantyla P, Pitkala KH. Changes in Institutionalized Older People's Dentition Status in Helsinki, 2003-2017. J Am Geriatr Soc. 2020 Jan;68(1):221-223. doi: 10.1111/jgs.16230. Epub 2019 Oct 26. No abstract available. PMID 31654530
- [Background] Saarela RKT, Hiltunen K, Kautiainen H, Roitto HM, Mantyla P, Pitkala KH. Oral hygiene and health-related quality of life in institutionalized older people. Eur Geriatr Med. 2022 Feb;13(1):213-220. doi: 10.1007/s41999-021-00547-8. Epub 2021 Jul 27. PMID 34313976
- [Background] Trujiilo K, Raisanen IT, Sorsa T, Patila T. Repeated Daily Use of Dual-Light Antibacterial Photodynamic Therapy in Periodontal Disease-A Case Report. Dent J (Basel). 2022 Sep 1;10(9):163. doi: 10.3390/dj10090163. PMID 36135158
- [Background] Suominen AL, Varsio S, Helminen S, Nordblad A, Lahti S, Knuuttila M. Dental and periodontal health in Finnish adults in 2000 and 2011. Acta Odontol Scand. 2018 Jul;76(5):305-313. doi: 10.1080/00016357.2018.1451653. Epub 2018 Mar 16. PMID 29546776
- See also: Berger, V., Bour, L., Carter, K. et al. A roadmap to using randomization in clinical trials. BMC Med Res Methodol 21, 168 (2021) — https://doi.org/10.1186/s12874-021-01303-z
- See also: Chan, AKY., Chu, CH., Ogawa, H., Hsiang-Hua Lai, E. Improving oral health of older adults for healthy ageing, Journal of Dental Sciences. (2023). ISSN 1991-7902 — https://doi.org/10.1016/j.jds.2023.10.018
- See also: Dodds, M., Roland, S., Edgar, M. et al. Saliva A review of its role in maintaining oral health and preventing dental disease. BDJ Team 2, 15123 (2015). — https://doi.org/10.1038/bdjteam.2015.123